CLINICAL TRIAL: NCT06354387
Title: A Pilot Study of Alectinib (Alecensa) in Combination with Nivolumab (Opdivo) in the Treatment of Recurrent or Refractory Hepatocellular Carcinoma Patients Guided with Serum Level of RNase1 and Tumor Expression of PD-L1
Brief Title: Alectinib in Combination with Nivolumab in the Treatment of Recurrent or Refractory HCC Patients Guided with Serum RNase1 and Tumor Expression of PD-L1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Fang Chiu, superintendent, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH110-REC3-246
Record Dates: First submitted 2024-03-18; First posted 2024-04-09 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — alectinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Experimental): open label
  Interventions: Drug: Alectinib (Alecensa), Nivolumab (Opdivo)

INTERVENTIONS:
Drug: Alectinib (Alecensa), Nivolumab (Opdivo) — Alectinib (Alecensa) in Combination with Nivolumab (Opdivo)
  Other Names: Alectinib (Alecensa)+ Nivolumab (Opdivo)

SUMMARY:
Hepatocellular carcinoma (HCC) is the fourth most common cause of cancer-related death and the second most deadly malignancy in Taiwan. Despite decades' intensive studies, surgery and local-regional chemo-embolization, radio-frequency ablation or radiation therapy remain the mainstay of HCC treatments.

DETAILED DESCRIPTION:
For HCC that are not resectable and not amenable to loco-regional therapies, the tyrosine kinase inhibitors (TKIs) sorafenib and its derivative regorafenib, lenvatinib and caboxantinib are of the standard systemic therapy. However, on average only marginal improvement of overall survival has been achieved with significant variation in response to TKI among patients. Effective predictive biomarkers to stratify patients for effective treatments have yet to be discovered.

In recent researches, the investigators have found RNase1 was highly expressed in nivolumab non-response HCC patients, and human ribonuclease1 (RNase1) secreted by tumor cells, was positive correlated with PD-L1 level in HCC patients. Notably, the investigators also found RNase1 regulates macrophage polarization and promotes immunosuppression in immunotherapy by activating ALK signaling in macrophage. the investigators showed that RNase1-overexpressing tumors were sensitive to ALK inhibitor and anti-PD-1 combinational therapy in HCC orthotopic mouse model.

Thus the investigators hypothesize that RNase1 is a potential biomarker for ALK inhibitor and anti-PD-1 combinational therapy in HCC. HCC patients who fit into the criteria would be benefit from ALK inhibitor (alectinib) and anti-PD-1 agent (nivolumab) combinational therapy. To test the role of circulatory RNase1 as a predictive biomarker for responsiveness to ALK inhibitor (alectinib) and anti-PD-1 agent (nivolumab) combinational therapy in Recurrent or Refractory HCC patients, the investigators propose the following pilot clinical studies in patients of HCC who failed the standard TKIs treatment. Total 8 evaluable subjects will be included. Participants will receive Alectinib (Alecensa) which has been approved for the treatment of ALK(+) NSCLC,ROS-1(+) NSCLC; and Nivolumab (Opdivo) has been approved for the treatment of several cancer types. Both of Alectinib and Nivolumab have also been under the reimbursement policy of Taiwan NHIA.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥20 years, at time of signing Informed Consent Form.
2. Histologically confirmed hepatocellular carcinoma, and the HCC cells harbor only wild-typed ALK.
3. Who has failed local treatments and at least one line of standard TKI treatment (sorafenib or lenvatinib) and not eligible for immune check point inhibitor treatment.
4. Life expectancy ≥ 12 weeks
5. At least one measurable (per RECIST 1.1) lesion. Patients who received prior local therapy (e.g., radiofrequency ablation or transarterial chemoembolization, etc.) are eligible provided the target lesion(s) have not been previously treated with local therapy or the target lesion(s) within the field of local therapy have subsequently progressed in accordance with RECIST version 1.1.
6. ECOG Performance Status of 0 or 1 within 7 days prior to registration
7. Child-Pugh class A (see Appendix) or B7-8 within 14 days prior to registration
8. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 7 days prior to registration, unless otherwise specified:

   1. ANC ≥ 1.5 *109/L(1500/μL) without granulocyte colony-stimulating factor support; platelet count ≥ 75*109/L(75000/μL) without transfusion; and hemoglobin≥ 90 g/L (9 g/dL)(patients may be transfused to meet this criterion).
   2. Liver transaminases (AST and ALT) ≤ 5 *upper limit of normal (ULN)
   3. Serum creatinine ≤ 1.5 * ULN or creatinine clearance≥ 50 mL/min (calculated using the Cockcroft-Gault formula)
   4. Urine dipstick for proteinuria ≤ 2+ (within 7 days prior to initiation of study treatment). Patients who have ≥ 2+ proteinuria on dipstick urinalysis at baseline will be eligible if he/she have daily protein excretion of ≤ 1g documented by a 24-hour urine collection.
9. Women of childbearing potential must agree to use contraceptive methods with a failure rate of < 1% per year (e.g., hormonal contraceptives that inhibit ovulation, copper intrauterine devices) during the treatment period and for at least 6 months after the last dose of Alectinib (Alecensa) in Combination with Nivolumab (Opdivo).
10. Men must agree to use contraceptive measures (condom plus an additional contraceptive method that together result in a failure rate of < 1% per year) during the treatment period and for 6 months after the last dose of Alectinib (Alecensa) in Combination with Nivolumab (Opdivo).

Exclusion Criteria:

1. Intolerant or severe allergic reactions to Alectinib (Alecensa) or Nivolumab (Opdivo)
2. Symptomatic central nervous system metastases. Brain metastases that have previously been treated and are stable for 4 weeks before the first dose date are allowed.
3. Prior treatment with Alectinib (Alecensa) and/or Nivolumab (Opdivo), or prior therapy with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody (or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways) for any reason.
4. Locoregional HCC therapy (e.g., TACE, RFA), systemic chemotherapy, hormonal therapy (e.g., tamoxifen) or investigational therapy within 4 weeks (or 5 half-lives, whichever is shorter) prior to Screening.
5. Life expectancy of less than 12 weeks
6. Major surgery or significant trauma within 14 days prior to Screening. Minor surgery within 7 days prior to Screening (excluding the placement of central/peripheral lines or skin biopsy).
7. Not recovered from the acute toxic effects of prior anticancer therapy, radiation or major surgery/significant trauma at Screening.
8. Major systemic diseases that the investigator considers inappropriate for participation
9. Known human immunodeficiency virus (HIV) infection
10. Concurrent active second malignancy for which the subject is receiving therapy, excluding non-melanomatous skin cancer, non-progressive prostate cancer treated with hormonal therapy, or carcinoma in situ of the cervix. Any cancer curatively treated >5 years prior to entry is permitted.
11. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection (e.g., tuberculosis) requiring antibiotic, antifungal, or antiviral therapy (other than antiHBV therapy), symptomatic heart failure, cardiac arrhythmia, acute or chronic pancreatitis or psychiatric illness/social situations that would limit compliance with study requirementsCNS metastasis.
12. Any active autoimmune disease or history of known autoimmune disease except for vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
13. Ongoing other concurrent investigational agents or anticancer therapy
14. Radiotherapy within 28 days prior to initiation of study treatment, except for palliative radiotherapy to bone lesions. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.
15. Presence of central nervous system (CNS) or leptomeningeal metastases. Patients with a history of CNS metastases are eligible for the study if he/she have received radiotherapy or surgery for the CNS metastases, and complete response (no evidence of residual CNS metastases) must be documented by brain CT scan at screening.
16. Requirement of systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
17. Prior organ allograft or allogeneic bone marrow transplantation.
18. Other severe acute or chronic medical or psychiatric conditions, or laboratory abnormality that may increase the risk associated with study participation and in the judgment of the investigator would make the patient inappropriate for entry into this study.
19. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX) are allowed

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | Baseline to EOT (up to 52 weeks)
  complete or partial response, as determined by the investigator according to RECIST v1.1

SECONDARY OUTCOMES:
PFS | Baseline to long term follow up (up to 52weeks)
  Progression-free survival

OTHER OUTCOMES:
TTP | Baseline to long term follow up (up to 52weeks)
  Time to tumor progression
DOR | Baseline to long term follow up (up to 52weeks)
  Duration of response
DCR | Baseline to long term follow up (up to 52weeks)
  Disease Control rate
OS | Baseline to long term follow up (up to 52weeks)
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Fang Chiu, Ph.D., Principal Investigator — China Medical University Hospital
Locations (1):
- CMUH, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No